CLINICAL TRIAL: NCT03338413
Title: Cognitive Rehabilitation in Patients With Active and Remitted Depression - a Randomized Controlled Trial
Brief Title: Cognitive Rehabilitation in Patients With Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: University of Oslo (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/666
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Depression
Keywords: Rehabilitation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal Management Training (Experimental)
  Interventions: Behavioral: Goal Management Training
- Computerized Cognitive Training (Experimental)
  Interventions: Behavioral: Computerized Cognitive Training

INTERVENTIONS:
Behavioral: Goal Management Training — 9 GMT modules will be administered in 9X2 hour sessions (ten groups). Manualized intervention; metacognitive strategies for improving attention and problem solving.
  Arms: Goal Management Training
Behavioral: Computerized Cognitive Training — 9 modules will be administered in 9x1 hour session (ten groups). Computerized Cognitive Training using commercially available web-based platforms based on neuroplasticity, developed to target skills such as attention, memory, speed of processing and executive functioning. Homework assignment between sessions.
  Other Names: Active control condition
  Arms: Computerized Cognitive Training

SUMMARY:
Depression is a highly prevalent and debilitating mental disorder, ranked one of the leading causes of disability worldwide. Several studies have identified neuropsychological deficits in populations of depressed patients affecting domains including attention, memory and executive functioning. These deficits often persist even in patients whose depressive symptoms have remitted. Cognitive impairment in depression represent a core feature of depression, and a valuable target for intervention. Identification of methods that would lead to amelioration would be of great clinical interest, and cognitive rehabilitation (CR) could be a potential way of achieving this. To date few studies on cognitive rehabilitation in depression has been conducted, but the preliminary results are promising. Still the demonstration of long-term effects and evidence relating to improved daily life executive functioning (i.e., generalization) is lacking. In the present study different group-based cognitive rehabilitation interventions will be compared. The aim of the study is to investigate if a group-based "brain training" intervention can improve executive function in patients with active and remitted depression. Efficacy will be assessed immediately after intervention, but also six months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Completed treatment for mild or moderate MDD
* Evidence of executive dysfunction in everyday life determined by (a) a structured interview or (b) a self-report Behavior Rating Inventory of Executive Function (BRIEF) T-score < 55.

Exclusion Criteria:

* Cognitive, sensory, physical, or language impairment affecting the capacity to complete the training program.
* Premorbid neurological disease or insult and/or comorbid neurological disorder.
* Reported ongoing alcohol or substance abuse.
* Psychotic disorders.
* Actively suicidal.
* Personality disorder sever enough to interfere with the protocol.
* Not fluent in Norwegian language.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Function (BRIEF: self and informant form) | Change from baseline up to 6 months
  Executive function in daily life (range:70-210). Higher score indicate greater executive dysfunction.

SECONDARY OUTCOMES:
Performance on Conners Continuous Performance test III incl. CATA | change from baseline up to 6 months
Performance on Wisconsin Card Sorting Test | change from baseline up to 6 months
Performance on D-KEFS Color Word Interference Test | change from baseline up to 6 months
Performance on The Emotional Stroop | change from baseline up to 6 months
Performance on the Emo 1-back task | change from baseline up to 6 months
Score on Cognitive Failures Questionnaire (CFQ) | change from baseline up to 6 months
  Assess frequency of cognitive failures (range:0-100). Higher Score indicate more frequent cognitive failures.
Score on Goal Attainment Scaling (GAS) | change from baseline up to 6 months
Score on Beck Depression Inventory II (BDI-II) | change from baseline up to 6 months
  Higher score indicate a higher level of depression (range: 0-63).
Score on Clinical Outcomes in Routine Evaluation Outcome Measure (CORE-OM) | change from baseline up to 6 months
  Assess the level of current psychological distress (range:0-136). Higher score indicate higher level of distress.
Score on General Perceived Self-Efficacy Scale | change from baseline up to 6 months
  Assess a general sense of perceived self-efficacy (range:10-40). Higher score indicate higher self-efficacy.
Score on Return to Work Self-Efficacy Scale (RTW-SE) | change from baseline up to 6 months
  Assess self-efficacy in the Return to work context (range:0-55). Higher score indicate higher self-efficacy.
Score on Difficulties in Emotion Regulation Scale (DERS) | change from baseline up to 6 months
  Higher score indicate a higher level of difficulties in emotion regulation (range:36-180).
Score on The Ruminative Response Scale (RRS) | change from baseline up to 6 months
  Higher score indicate a higher level of ruminative responses (range: 22-88).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Joner, Study Director — Lovisenberg Diaconal Hospital
Locations (1):
- Lovisenberg Diaconal Hospital, Oslo, Norway